CLINICAL TRIAL: NCT01960660
Title: A Marketing-oriented Study to Evaluate the Comparative Bioavailability of Omega-3 Fatty Acids From Four Different Natural Health Products
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nordic Pharma, USA (Industry)
Collaborators: Nutrasource Pharmaceutical and Nutraceutical Services, Inc. (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 12.0216; 12-03-001 (Other: Canadian SHIELD Ethics Review Board)
Record Dates: First submitted 2013-10-08; First posted 2013-10-10 (Estimated); Last update posted 2015-12-14 (Estimated); Status verified 2015-12

CONDITIONS: Comparative Bioavailability
Keywords: Fish Oil; EPA; DHA; Omega-Score; Lipemic Index; ethyl esters; triglycerides; phospholipids
MeSH Terms: conditions — Hyperlipidemias | interventions — Fatty Acids, Omega-3; Docosahexaenoic Acids

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Investigational Product (Experimental): Omega-3 fatty acids in the form of triglycerides
  Interventions: Dietary Supplement: Omega-3 Fatty Acids
- Comparator Product 1 (Active Comparator): Omega-3 fatty acids in the form of ethyl esters.
  Interventions: Dietary Supplement: Omega-3 Fatty Acids
- Comparator Product 2 (Active Comparator): Omega-3 fatty acids in the form of phospholipids from krill oil.
  Interventions: Dietary Supplement: Omega-3 Fatty Acids
- Comparator Product 3 (Active Comparator): Omega-3 fatty acids from salmon oil.
  Interventions: Dietary Supplement: Omega-3 Fatty Acids

INTERVENTIONS:
Dietary Supplement: Omega-3 Fatty Acids
  Other Names: EPA: Eicosapentaenoic acid (20:5(n-3)); DHA: Docosahexaenoic acid (22:6(n-3))

SUMMARY:
Supplementation with omega-3 fatty acids has been extensively researched and is known to provide healthful benefits for patients with a diversity of conditions and diseases. Not all omega-3 supplements are created equally however; some sources of omega-3 fatty acids are superior to others due to a greater bioavailability of omega-3 fatty acids than others, differences in source material, and processing techniques.

The purpose of this study is to determine which marketed omega-3 product provided the greatest effect, as measured against its' label claim and recommended dosage.

ELIGIBILITY:
Inclusion Criteria:

* Participant is fluent in English
* Participant understands the study requirements and is willing to comply with the protocol
* Participant is willing to provide written informed consent
* Participant is 18 years of age or older

Exclusion Criteria:

* Unwilling or unable to provide written consent
* Participant has taken omega-3 supplements in the last 3 months
* Participants consumes fish on a regular basis (more than 1 serving per week)
* Females who are pregnant or breastfeeding
* Participant has an allergy to fish or seafood
* Participant has been diagnosed with any medical illness or conditions
* Participant has a history of drug dependence or substance abuse (excluding nicotine)
* Participant is taking cholesterol or triglyceride lowering medications or supplements (statins, niacin, carnitine, fibrates)
* Individual has difficulty giving multiple blood samples

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2012-05; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Omega-Score | Change from Baseline in Omega-Score at 28 days
  The Omega ScoreTM is a measurement of the levels of the Omega-3 Fatty Acids in a blood sample. The summed amounts of these Omega-3 Fatty Acids (EPA+DPA+DHA) as a % of the total fatty acids represents the Omega ScoreTM in whole blood.

SECONDARY OUTCOMES:
Lipemic IndexTM | Change from Baseline in Lipemic Index at 28 days
  The Lipemic Index™ is the post-prandial rise in TG levels over a 5-hour period, following the consumption drink containing a measured amount of fat, carbohydrate and protein.

CONTACTS AND LOCATIONS:
Overall Officials: Maggie D Laidlaw, Ph.D, Principal Investigator — Nutrasource Diagnostics; Carla Cockerline, M.Sc, Study Director — Nutrasource Diagnostics
Locations (1):
- Nutrasource Diagnostics Inc, Guelph, Ontario, Canada

REFERENCES:
- [Derived] Laidlaw M, Cockerline CA, Rowe WJ. A randomized clinical trial to determine the efficacy of manufacturers' recommended doses of omega-3 fatty acids from different sources in facilitating cardiovascular disease risk reduction. Lipids Health Dis. 2014 Jun 21;13:99. doi: 10.1186/1476-511X-13-99. PMID 24952576